CLINICAL TRIAL: NCT05229263
Title: Exploratory Multicentre Clinical Study to Assess Repeatibility, Reproducibility, Acceptability and Clinical Validity of Multiparametric Renal Magnetic Resonance Imaging
Brief Title: Multiparametric MRI in Healthy Volunteers and CKD Patients
Acronym: RESPECT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Clinica Universidad de Navarra, Universidad de Navarra (Other); Aarhus University Hospital (Other); Heidelberg University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RESPECT
Record Dates: First submitted 2022-01-14; First posted 2022-02-08 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Diseases; Healthy
Keywords: Multiparametric MRI; Chronic kidney disease; Standardization; Clinical validity
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Two groups of subjects (healthy volunteers and CKD patients) are involved in the study and will follow separate workflows.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy volunteers (Experimental)
  Interventions: Diagnostic Test: Non- contrast Enhanced Multiparametric Renal Magnetic Resonance
- CKD patients (Experimental)
  Interventions: Diagnostic Test: Non- contrast Enhanced Multiparametric Renal Magnetic Resonance

INTERVENTIONS:
Diagnostic Test: Non- contrast Enhanced Multiparametric Renal Magnetic Resonance — MRI is performed in a single multiparametric scan session with no need for contrast agents, and to depict changes in tissue microstructure associated with inflammation and fibrosis plus alterations in oxygenation.

SUMMARY:
Chronic kidney disease (CKD) is a global health concern because more than 10% of the world's population have it, its prevalence is increasing, and CKD is an important contributor to morbidity and mortality for this population.

The majority of the people with CKD aren't aware and there are not available tools for early CKD detection and for an accurate prediction on these patients. Many CKD patients exhibit progressive renal dysfunction, demonstrating a failure of current, non-specific therapeutic strategies. Better methods are urgently needed for i) early diagnosis of CKD, and prediction of its progression for improved stratification of patients and better targeting of current treatments; and ii) to directly assess structural and functional responses of the kidney to new therapies and identify those patients who respond.

Over the past decade, renal Magnetic Resonance Imaging (MRI) has emerged as a promising technique for improved understanding and characterisation of renal pathophysiology. Compared to histopathology, MRI is non-invasive and avoids sampling bias by characterising the entire kidney with high spatial resolution.

In spite of a number of single centre studies showing renal MRI feasibility and potential to address a number of key clinical questions, current methodological differences across studies hinder reliable comparisons of the results, which can only be regarded as preliminary. Standardization of acquisition and processing protocols across centres is therefore needed, and this will also lead to the possibility to provide preliminary data of the multiparametric renal MRI clinical validity and utility.

The purpose of this study is to standardize, assess the feasibility and provide preliminary evidence of clinical validity and utility of the multiparametric renal MRI.

To reach this goal two groups of subjects are involved:

* Group 1 (healthy volunteers). In this group the repeatibility and reproducibility of multiparametric renal MRI will be assessed.
* Group 2 (CKD patients). In this group the feasibility, the acceptability, the reproducibility and the preliminary clinical validity of multiparametric renal MRI will be assessed.

ELIGIBILITY:
Inclusion Criteria:

GROUP 1:

1. Provision of written informed consent prior to any study specific procedures
2. Male and female subjects aged more than18 years
3. Normotensive (office Systolic Blood Pressure values < 140 mmHg and Diastolic Blood Pressure values ≤ 90 mmHg)
4. Normal renal condition for age (established by estimating Glomerular Filtration Rate using CKD-EPI, Chronic Kidney Disease Epidemiology Collaboration, Creatinine Equation)
5. Negative result upon urine dipstick testing for haematuria or proteinuria.
6. Normal Urine Albumin-to-Creatinine Ratio (UACR) (<30 mg/g)

GROUP 2:

1. Provision of written informed consent prior to any study specific procedures
2. Male and female patients aged more than18 years
3. CKD stage 2 or 3, with albuminuria up to 2000 mg

Exclusion Criteria:

GROUP 1 and 2

1. Previous enrollment in the present study
2. Contraindications to MRI including due to:

   * Claustrophobia
   * Pregnancy
   * Cardiac pacemakers or other MRI-incompatible prostheses

Only GROUP 2:

1. Urine Albumin-to-Creatinine Ratio higher than 2000 mg/g or 24h urine total albumin >2 g
2. Polycystic kidney disease, renovascular disease, active/current nephrotic syndrome, reflux nephropathy and known congenital renal diseases or solitary kidney.
3. Active malignancy or acute or chronic inflammatory disease, HIV
4. Acute kidney injury, as defined by the the KDIGO guidelines, during the last three months.
5. Need of a new immunosuppressive therapy for treating renal disease relapse in the preceding three months.
6. Dialysis or kidney transplantation
7. CKD stages 4 or 5
8. New medication in the preceding two weeks (diuretic, hypertensive, SGLT2 treatment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-11-25 (Actual); Primary Completion 2025-03-13 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
GROUP 1: within subject total kidney volume coefficient of variation in few hour time | At day 0
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated in few hour time to assess total kidney volume repeatability in the whole group of healthy volunteers
GROUP 1: within subject total kidney volume coefficient of variation after 1-2 weeks | At day 7-14
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated after 1-2 weeks to assess total kidney volume reproducibility in the whole group of healthy volunteers
GROUP 1: within subject renal artery blood flow coefficient of variation in few hour time | At day 0
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated in few hour time to assess renal artery blood flow repeatability in the whole group of healthy volunteers
GROUP 1: within subject renal artery blood flow coefficient of variation after 1-2 weeks | At day 7-14
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated after 1-2 weeks to assess renal artery blood flow reproducibility in the whole group of healthy volunteers
GROUP 1: within subject cortical perfusion coefficient of variation in few hour time | At day 0
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated in few hour time to assess cortical perfusion repeatability in the whole group of healthy volunteers
GROUP 1: within subject cortical perfusion coefficient of variation after 1-2 weeks | At day 7-14
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated after 1-2 weeks to assess cortical perfusion reproducibility in the whole group of healthy volunteers
GROUP 1: within subject cortical and medullary T1 coefficient of variation in few hour time | At day 0
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated in few hour time to assess cortical and medullary T1 repeatability in the whole group of healthy volunteers
GROUP 1: within subject cortical and medullary T1 coefficient of variation after 1-2 weeks | At day 7-14
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated after 1-2 weeks to assess cortical and medullary T1 reproducibility in the whole group of healthy volunteers
GROUP 1: within subject cortical and medullary T2 coefficient of variation in few hour time | At day 0
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated in few hour time to assess cortical and medullary T2 repeatability in the whole group of healthy volunteers
GROUP 1: within subject cortical and medullary T2 coefficient of variation after 1-2 weeks | At day 7-14
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated after 1-2 weeks to assess cortical and medullary T2 reproducibility in the whole group of healthy volunteers
GROUP 1: within subject cortical and medullary R2* coefficient of variation in few hour time | At day 0
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated in few hour time to assess cortical and medullary R2* repeatability in the whole group of healthy volunteers
GROUP 1: within subject cortical and medullary R2* coefficient of variation after 1-2 weeks | At day 7-14
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated after 1-2 weeks to assess cortical and medullary R2* reproducibility in the whole group of healthy volunteers
GROUP 1: within subject cortical and medullary ADC coefficient of variation in few hour time | At day 0
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated in few hour time to assess cortical and medullary ADC repeatability in the whole group of healthy volunteers
GROUP 1: within subject cortical and medullary ADC coefficient of variation after 1-2 weeks | At day 7-14
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated after 1-2 weeks to assess cortical and medullary ADC reproducibility in the whole group of healthy volunteers
GROUP 2 - Percentage of complete renal MRI data collection and analysis | At day 0
  Percentage of complete renal MRI data acquired and generated by MRI data processing in the whole group of CKD patients, to assess feasibility of multiparametric renal MRI in CKD patients

SECONDARY OUTCOMES:
GROUP 1 - within subject renal total kidney volume coefficient of variation in few hour time by gender | At day 0
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated in few hour time in male and female healthy volunteers to assess differences in total kidney volume repeatability between genders
GROUP 1 - within subject renal artery blood flow coefficient of variation in few hour time by gender | At day 0
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated in few hour time in male and female healthy volunteers to assess differences in renal artery blood flow repeatability between genders
GROUP 1 - within subject cortical perfusion coefficient of variation in few hour time by gender | At day 0
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated in few hour time in male and female healthy volunteers to assess differences in cortical perfusion repeatability between genders
GROUP 1 - within subject cortical and medullary T1 coefficient of variation in few hour time by gender | At day 0
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated in few hour time in male and female healthy volunteers to assess differences in cortical and medullary T1 repeatability between genders
GROUP 1 - within subject cortical and medullary T2 coefficient of variation in few hour time by gender | At day 0
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated in few hour time in male and female healthy volunteers to assess differences in cortical and medullary T2 repeatability between genders
GROUP 1 - within subject cortical and medullary R2* coefficient of variation in few hour time by gender | At day 0
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated in few hour time in male and female healthy volunteers to assess differences in cortical and medullary R2* repeatability between genders
GROUP 1 - within subject cortical and medullary ADC coefficient of variation in few hour time by gender | At day 0
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated in few hour time in male and female healthy volunteers to assess differences in cortical and medullary ADC repeatability between genders
GROUP 1 - within subject total kidney volume coefficient of variation in few hour time by age | At day 0
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated in few hour time in healthy volunteers of different age to assess differences in total kidney volume repeatability between age classes
GROUP 1 - within subject renal artery blood flow coefficient of variation in few hour time by age | At day 0
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated in few hour time in healthy volunteers of different age to assess difference in renal artery blood flow repeatability between age classes
GROUP 1 - within subject cortical perfusion coefficient of variation in few hour time by age | At day 0
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated in few hour time in healthy volunteers of different age to assess differences in cortical perfusion repeatability between age classes
GROUP 1 - within subject cortical and medullary T1 coefficient of variation in few hour time by age | At day 0
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated in few hour time in healthy volunteers of different age to assess differences in cortical and medullary T1 repeatability between age classes
GROUP 1 - within subject cortical and medullary T2 coefficient of variation in few hour time by age | At day 0
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated in few hour time in healthy volunteers of different age to assess differences in cortical and medullary T2 repeatability between age classes
GROUP 1 - within subject cortical and medullary R2* coefficient of variation in few hour time by age | At day 0
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated in few hour time in healthy volunteers of different age to assess differences in cortical and medullary R2* repeatability between age classes
GROUP 1 - within subject cortical and medullary ADC coefficient of variation in few hour time by age | At day 0
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated in few hour time in healthy volunteers of different age to assess differences in cortical and medullary ADC repeatability between age classes
GROUP 1 - within subject total kidney volume coefficient of variation after 1-2 weeks by gender | At day 7-14
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated after 1-2 weeks in male and female healthy volunteers to assess differences in total kidney volume reproducibility between genders
GROUP 1 - within subject renal artery blood flow coefficient of variation after 1-2 weeks by gender | At day 7-14
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated after 1-2 weeks in male and female healthy volunteers to assess differences in renal artery blood flow reproducibility between genders
GROUP 1 - within subject cortical perfusion coefficient of variation after 1-2 weeks by gender | At day 7-14
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated after 1-2 weeks in male and female healthy volunteers to assess differences in cortical perfusion reproducibility between genders
GROUP 1 - within subject cortical and medullary T1 coefficient of variation after 1-2 weeks by gender | At day 7-14
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated after 1-2 weeks in male and female healthy volunteers to assess difference in cortical and medullary T1 reproducibility between genders
GROUP 1 - within subject cortical and medullary T2 coefficient of variation after 1-2 weeks by gender | At day 7-14
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated after 1-2 weeks in male and female healthy volunteers to assess differences in cortical and medullary T2 reproducibility between genders
GROUP 1 - within subject cortical and medullary R2* coefficient of variation after 1-2 weeks by gender | At day 7-14
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated after 1-2 weeks in male and female healthy volunteers to assess differences in cortical and medullary R2* reproducibility between genders
GROUP 1 - within subject cortical and medullary ADC coefficient of variation after 1-2 weeks by gender | At day 7-14
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated after 1-2 weeks in male and female healthy volunteers to assess differences in cortical and medullary ADC reproducibility between genders
GROUP 1 - within subject total kidney volume coefficient of variation after 1-2 weeks by age | At day 7-14
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated after 1-2 weeks in healthy volunteers of different age to assess differences in total kidney volume reproducibility between age classes
GROUP 1 - within subject renal artery blood flow coefficient of variation after 1-2 weeks by age | At day 7-14
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated after 1-2 weeks in healthy volunteers of different age to assess differences in renal artery blood flow reproducibility between age classes
GROUP 1 - within subject cortical perfusion coefficient of variation after 1-2 weeks by age | At day 7-14
  Within subject coefficient of variation of measures computed by multiparametric renal MRI after 1-2 weeks in healthy volunteers of different age to assess differences in cortical perfusion reproducibility between age classes
GROUP 1 - within subject cortical and medullary T1 coefficient of variation after 1-2 weeks by age | At day 7-14
  Within subject coefficient of variation of measures computed by multiparametric renal MRI after 1-2 weeks in healthy volunteers of different age to assess differences in cortical and medullary T1 reproducibility between age classes
GROUP 1 - within subject cortical and medullary T2 coefficient of variation after 1-2 weeks by age | At day 7-14
  Within subject coefficient of variation of measures computed by multiparametric renal MRI after 1-2 weeks in healthy volunteers of different age to assess differences in cortical and medullary T2 reproducibility between age classes
GROUP 1 - within subject cortical and medullary R2* coefficient of variation after 1-2 weeks by age | At day 7-14
  Within subject coefficient of variation of measures computed by multiparametric renal MRI after 1-2 weeks in healthy volunteers of different age to assess differences in cortical and medullary R2* reproducibility between age classes
GROUP 1 - within subject cortical and medullary ADC coefficient of variation after 1-2 weeks by age | At day 7-14
  Within subject coefficient of variation of measures computed by multiparametric renal MRI after 1-2 weeks in healthy volunteers of different age to assess differences in cortical and medullary ADC reproducibility between age classes
GROUP 1 - Multiparametric MRI acceptability in healthy volunteers. | At day 0
  Multiparametric MRI acceptability, in terms of comfort level and degree of satisfaction, assessed by a specific 9-item questionnaire ([9-45] range of values, with highest values denoting highest acceptability [Chen S, et al. J Appl Clin Med Phys. 2019; 20(7):184-192]) in healthy volunteers.
GROUP 2 - Multiparametric MRI acceptability in CKD patients. | At day 0
  Multiparametric MRI acceptability, in terms of comfort level and degree of satisfaction, assessed by a specific 9-item questionnaire ([9-45] range of values, with highest values denoting highest acceptability [Chen S, et al. J Appl Clin Med Phys. 2019; 20(7):184-192]) in CKD patients.
GROUP 2 - within subject total kidney volume coefficient of variation after 1-2 weeks | At day 7-14
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated after 1-2 weeks to assess total kidney volume reproducibility in CKD patients
GROUP 2 - within subject renal artery blood flow coefficient of variation after 1-2 weeks | At day 7-14
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated after 1-2 weeks to assess renal artery blood flow reproducibility in CKD patients
GROUP 2 - within subject cortical perfusion coefficient of variation after 1-2 weeks | At day 7-14
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated after 1-2 weeks to assess cortical perfusion reproducibility in CKD patients
GROUP 2 - within subject cortical and medullary T1 coefficient of variation after 1-2 weeks | At day 7-14
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated after 1-2 weeks to assess cortical and medullary T1 reproducibility in CKD patients
GROUP 2 - within subject cortical and medullary T2 coefficient of variation after 1-2 weeks | At day 7-14
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated after 1-2 weeks to assess cortical and medullary T2 reproducibility in CKD patients
GROUP 2 - within subject cortical and medullary R2* coefficient of variation after 1-2 weeks | At day 7-14
  Within subject coefficient of variation of measures computed by multiparametric renal MR repeated after 1-2 weeks to assess cortical and medullary R2* reproducibility in CKD patients
GROUP 2 - within subject cortical and medullary ADC coefficient of variation after 1-2 weeks | At day 7-14
  Within subject coefficient of variation of measures computed by multiparametric renal MRI repeated after 1-2 weeks to assess cortical and medullary ADC reproducibility in CKD patients
GROUP 2 - Correlation coefficient between MRI-based parameters and eGFR | At day 0
  Assessment of the correlation coefficient between MRI-based parameters and eGFR to provide preliminary evidence of the nature and degree of change in multiparametric MRI measures across different stages of CKD

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Remuzzi, MD, Study Chair — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (4):
- Aarhus University Hospital, Department of Renal Medicine, Århus N, Århus N, Denmark
- University Medical Center Mannheim, Medical Faculty Mannheim, Heidelberg University, Heidelberg, Mannheim, Germany
- Centro di Ricerche Cliniche per le Malattie Rare "Aldo e Cele Daccò", Ranica, BG, Italy
- Clínica Universidad de Navarra, Pamplona, Navarre, Spain